CLINICAL TRIAL: NCT03484091
Title: Comparison of Single Intra-articular Injection of Hyruan-One With Hylan G-F 20 in Knee Osteoarthritis: A Randomized Double-blind, Saline-controlled Trial
Brief Title: Comparison of Single Intra-articular Injection of Hyruan-One With Hylan G-F 20 in Knee Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Supakit Kanitnate, Department of orthopaedics, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OrthoTU09
Record Dates: First submitted 2018-02-24; First posted 2018-03-30 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2018-03

CONDITIONS: Knee Osteoarthritis
Keywords: Hyruan-One; Hylan G-F 20; Hyaluronic acid; Knee osteoarthritis; Pain level
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — hylan; Saline Solution

STUDY DESIGN:
Intervention Model Description: A double-blind, placebo controlled RCT
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- H group (Experimental): Single dose of Hyruan-One 3 mL intra-articular knee injection.
  Interventions: Drug: Hyruan-One
- S group (Active Comparator): Single dose of Hylan G-F 20 (Synvisc) 6 mL intra-articular knee injection.
  Interventions: Drug: Hylan G-F 20
- N group (Placebo Comparator): Single dose of normal saline 6 mL intra-articular knee injection.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Hyruan-One — single dose intra-articular injection
  Arms: H group
Drug: Hylan G-F 20 — single dose intra-articular injection
  Other Names: Synvisc
  Arms: S group
Drug: Normal saline — single dose intra-articular injection
  Arms: N group

SUMMARY:
We compare the efficacy of intra-articular injection of Hyruan-One with Hylan G-F 20 and placebo (NSS) controlled in a double-blind RCT.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic primary knee osteoarthritis with failed conservative treatment for at least 3 months
* Gave informed consent
* Can do questionnaires

Exclusion Criteria:

* Severe deformity (varus or valgus from a mechanical axis more than 10 degrees
* Allergy to hyaluronic acid
* Pain in the hip or ankle
* Post-traumatic or post surgery of lower extremity
* Post-infection of the knee
* Previous hyaluronic acid injection within 6 months
* Pregnancy or lactation
* Underlying Rheumatoid arthritis, stroke, malignancy, venous occlusion

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Pain level | 6 months after injection
  visual analog scale for pain (0-100) in between groups
Change from pre-injection pain level at 6 months | 6 months
  compare visual analog scale for pain (0-100) between pre-injection and post-injection

SECONDARY OUTCOMES:
pain level in any time pints | post-injection 1, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24 weeks
  visual analog scale for pain (0-100)
Modified WOMAC | post-injection 2 weeks, 1, 2, 3,4, 5, 6 months
  measure modified WOMAC score (0-96)
Lequesne index | post-injection 2 weeks, 1, 2, 3,4, 5, 6 months
  measure Lequesne index for knee osteoarthritis (4-24)
SF-36 | post-injection 2 weeks, 1, 2, 3,4, 5, 6 months
  measure short from health survey 36 items
Time up and go test | post-injection 1, 3, 6 months
  recorded time Up and Go test (minutes)
Complications | post-injection 1, 2 weeks
  assess complications after injection by phone

CONTACTS AND LOCATIONS:
Overall Officials: Nattapol Tammachote, MD, Principal Investigator — Thammasat University
Locations (1):
- Thammasat University, Khlong Luang, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: Undecided